CLINICAL TRIAL: NCT01592370
Title: Multiple Phase 1/2 Cohorts of Nivolumab Monotherapy or Nivolumab Combination Regimens Across Relapsed/Refractory Hematologic Malignancies
Brief Title: An Investigational Immuno-Therapy Study to Determine the Safety and Effectiveness of Nivolumab and Daratumumab in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-039; 2018-001030-17 (EudraCT Number)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2022-02-17 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma | interventions — Nivolumab; Ipilimumab; lirilumab; daratumumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Nivolumab monotherapy (Dose Escalation) (Experimental): Nivolumab solution intravenously as specified
  Non-randomized
  Enrollment is closed for this cohort
  Interventions: Biological: Nivolumab
- Nivolumab + Ipilimumab (Experimental): Nivolumab and Ipilimumab solution intravenously as specified
  Non-randomized
  Enrollment is closed for this cohort
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab + Lirilumab (Experimental): Non-randomized
  Nivolumab: 3 mg/kg given every 2 weeks Lirilumab: 3 mg/kg given every 4 weeks
  Enrollment is closed for this cohort
  Interventions: Biological: Nivolumab; Biological: Lirilumab
- Nivo + Dara + Pom + Dexa vs. Nivo + Dara (Experimental): Randomized
  Nivolumab:
  Cycle 1: 240 mg Day 15 Cycle 2-6: 240 mg Days 1, 15 Cycle 7 & beyond: 480 mg Day 1
  Daratumumab:
  Cycle 1-2: 16 mg/kg Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg Days 1, 15 Cycle 7 & beyond: 16 mg/kg Day 1
  Pomalidomide:
  4 mg po (by mouth) daily on Days 1 - 21 of each 28-day cycle
  Dexamethasone:
  Weeks without daratumumab dosing:
  * 40 mg po daily (Days 1, 8, 15, 22) of each 28-day cycle for participants ≤ 75 years old
  * 20 mg po daily (Days 1, 8, 15, 22) of each 28-day cycle for participants > 75 years old
  Weeks with daratumumab dosing:
  * 20 mg iv before the daratumumab infusion and 20 mg po after the daratumumab infusion in participants ≤ 75 years old
  * 16 mg iv before the daratumumab infusion and 4 mg po after the daratumumab infusion in participants > 75 years old
  Enrollment is closed for this cohort
  Interventions: Biological: Nivolumab; Biological: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone
- Daratumumab vs. Nivolumab + Daratumumab (Experimental): Randomized
  Nivolumab:
  Cycle 1: 240 mg Day 15 Cycle 2 & beyond: 480 mg Day 1
  Daratumumab:
  Cycle 1-2: 16 mg/kg Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg Days 1, 15 Cycle 7 & beyond: 16 mg/kg Day 1
  Interventions: Biological: Nivolumab; Biological: Daratumumab

INTERVENTIONS:
Biological: Nivolumab — Administered by intravenous (IV) infusion
  Other Names: BMS-936558; Opdivo
Biological: Ipilimumab — Administered by IV infusion
  Other Names: Yervoy; BMS-734016; MDX010
  Arms: Nivolumab + Ipilimumab
Biological: Lirilumab — Administered by IV infusion
  Other Names: BMS-986015
  Arms: Nivolumab + Lirilumab
Biological: Daratumumab — Administered by IV infusion
  Other Names: Darzalex
  Arms: Daratumumab vs. Nivolumab + Daratumumab; Nivo + Dara + Pom + Dexa vs. Nivo + Dara
Drug: Pomalidomide — Administered PO
  Other Names: Pomalyst
  Arms: Nivo + Dara + Pom + Dexa vs. Nivo + Dara
Drug: Dexamethasone — Administered PO and by IV infusion
  Other Names: Intensol
  Arms: Nivo + Dara + Pom + Dexa vs. Nivo + Dara

SUMMARY:
The purpose of this study is to determine the side effects of treatment of the combination of nivolumab and daratumumab in participants with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
NOTE: Currently, this study is only open to nivolumab+daratumumab vs daratumumab monotherapy in multiple myeloma patients.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Have received at least 3 prior lines of therapy, including a proteasome inhibitor [PI] and an immunomodulatory agent [IMiD] OR have disease that is double refractory to a PI and IMiD
* More than 12 weeks post-transplant of your own blood forming stem cells (autologous transplant)
* Have detectable disease measured by a specific protein in your blood and/or urine
* Must consent to bone marrow aspirate or biopsy.

Exclusion Criteria:

* Solitary bone or extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia, or monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), primary amyloidosis, Waldenstrom's macroglobulinemia, POEMS syndrome or active plasma cell leukemia
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti CTLA 4, or anti-CD38 antibody, or allogeneic stem cell transplantation
* Seropositive for human immunodeficiency virus (HIV), Hepatitis B surface antigen or Hepatitis C antibody positive (except if HCV-RNA negative), or history of active chronic hepatitis B or C
* History of central nervous system involvement or symptoms suggestive of central nervous system involvement by multiple myeloma

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-08-02 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (43):
- United States (32):
  - Local Institution - 0035, Clovis, California
  - Division Of Hematology & Oncology Ctr. For Health Sciences, Los Angeles, California
  - Local Institution - 0012, Los Angeles, California
  - Local Institution - 0017, Aurora, Colorado
  - Local Institution - 013, New Haven, Connecticut
  - Local Institution - 0023, Orlando, Florida
  - Local Institution - 0037, Skokie, Illinois
  - Local Institution - 0019, Indianapolis, Indiana
  - Local Institution - 0018, Westwood, Kansas
  - Local Institution - 0003, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 0009, Boston, Massachusetts
  - Local Institution - 0015, Boston, Massachusetts
  - Local Institution - 0011, Ann Arbor, Michigan
  - University Of Michigan Health System, Ann Arbor, Michigan
  - Local Institution - 0002, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Local Institution - 0033, Omaha, Nebraska
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Local Institution - 0014, Hackensack, New Jersey
  - Local Institution - 0001, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 0028, Columbus, Ohio
  - Local Institution - 0006, Portland, Oregon
  - OHSU Center for Hematologic Malignancies, Portland, Oregon
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 0007, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 0004, Philadelphia, Pennsylvania
  - Huntsman Cancer Institute At The Univ. Of Utah, Salt Lake City, Utah
  - Local Institution - 0005, Salt Lake City, Utah
- Belgium (3):
  - Local Institution - 0045, Ghent
  - Local Institution - 0047, Sint-Niklaas
  - Local Institution, Yvoir
- France (2):
  - Local Institution - 0043, Poitiers, Vienne
  - Local Institution - 0044, Nantes
- Local Institution - 0039, Athens, Greece
- Local Institution, Bologna, Italy
- Poland (4):
  - Local Institution, Chorzów
  - Local Institution - 0040, Poznan
  - Local Institution - 0049, Warsaw
  - Local Institution - 0042, Wroclaw

REFERENCES:
- [Derived] Lesokhin AM, Ansell SM, Armand P, Scott EC, Halwani A, Gutierrez M, Millenson MM, Cohen AD, Schuster SJ, Lebovic D, Dhodapkar M, Avigan D, Chapuy B, Ligon AH, Freeman GJ, Rodig SJ, Cattry D, Zhu L, Grosso JF, Bradley Garelik MB, Shipp MA, Borrello I, Timmerman J. Nivolumab in Patients With Relapsed or Refractory Hematologic Malignancy: Preliminary Results of a Phase Ib Study. J Clin Oncol. 2016 Aug 10;34(23):2698-704. doi: 10.1200/JCO.2015.65.9789. Epub 2016 Jun 6. PMID 27269947
- [Derived] Ansell SM, Lesokhin AM, Borrello I, Halwani A, Scott EC, Gutierrez M, Schuster SJ, Millenson MM, Cattry D, Freeman GJ, Rodig SJ, Chapuy B, Ligon AH, Zhu L, Grosso JF, Kim SY, Timmerman JM, Shipp MA, Armand P. PD-1 blockade with nivolumab in relapsed or refractory Hodgkin's lymphoma. N Engl J Med. 2015 Jan 22;372(4):311-9. doi: 10.1056/NEJMoa1411087. Epub 2014 Dec 6. PMID 25482239
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the phase 1 nivo monotherapy dose escalation included in this study, it was derived from CA209-003. It was concluded that 3mg/kg of nivolumab would be used for the dose expansion phase 2 of this study (CA209-039) based on the conclusions derived from CA209-003.
Pre-assignment Details: 316 participants treated
Groups:
- Nivolumab Monotherapy (Expansion): 3mg/kg of nivolumab
- Nivolumab + Ipilimumab: 3 mg/kg of nivolumab and
  1 mg/kg of ipilimumab Q3W for 4 doses, followed by nivolumab alone at 3 mg/kg Q2W
- Nivolumab + Lirilumab: 3 mg/kg of nivolumab Q2W + 3 mg/kg of lirilumab Q4W
- Nivolumab + Daratumumab_Cohort A1: ND regimen: Nivolumab (240 mg up to cycle 6, then 480 mg) + Daratumumab (16 mg/Kg)
- Nivolumab + Daratumumab_Cohort A2: ND-PD regimen; Nivolumab + Daratumumab + Pomalidomide + Dexamethasone
- Nivolumab + Daratumumab_Cohort B1: ND regimen: Nivolumab (240 mg cycle 1, then 480 mg) + Daratumumab (16 mg/Kg)
- Nivolumab + Daratumumab_Cohort B2: D regimen: Daratumumab alone
Period: Overall Study
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab | Nivolumab + Daratumumab_Cohort A1 | Nivolumab + Daratumumab_Cohort A2 | Nivolumab + Daratumumab_Cohort B1 | Nivolumab + Daratumumab_Cohort B2
Started (= Number of participants randomized) | 105 | 65 | 72 | 6 | 7 | 43 | 22
Completed | 1 | 40 | 0 | 1 | 1 | 7 | 6
Not Completed | 104 | 25 | 72 | 5 | 6 | 36 | 16
Not completed — Disease Progression | 62 | 16 | 52 | 3 | 3 | 31 | 14
Not completed — Study Drug Toxicity | 14 | 3 | 0 | 0 | 0 | 0 | 1
Not completed — AE unrelated to study drug | 4 | 3 | 0 | 0 | 0 | 0 | 1
Not completed — Request to discontinue study treatment | 5 | 0 | 2 | 0 | 1 | 2 | 0
Not completed — Withdrew consent | 1 | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 11 | 1 | 7 | 1 | 0 | 0 | 0
Not completed — No longer meets study criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Reasons | 6 | 0 | 10 | 0 | 0 | 1 | 0
Not completed — Not Treated | 0 | 0 | 0 | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab | Nivolumab + Daratumumab_Cohort A1 | Nivolumab + Daratumumab_Cohort A2 | Nivolumab + Daratumumab_Cohort B1 | Nivolumab + Daratumumab_Cohort B2 | Total
Number analyzed (Participants) | 105 | 65 | 72 | 6 | 7 | 43 | 22 | 320
Age, Categorical [Count of Participants; unit: Participants] — Population: All treated participants for Nivo mono, Nivo + Ipi , Nivo + Liri and all randomized participants for Nivo Dara
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 66 | 46 | 52 | 3 | 3 | 17 | 11 | 198
    >=65 years | 39 | 19 | 20 | 3 | 4 | 26 | 11 | 122
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants for Nivo mono, Nivo + Ipi , Nivo + Liri and all randomized participants for Nivo Dara
  Participants
    Female | 45 | 28 | 26 | 3 | 3 | 25 | 8 | 138
    Male | 60 | 37 | 46 | 3 | 4 | 18 | 14 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants for Nivo mono, Nivo + Ipi , Nivo + Liri and all randomized participants for Nivo Dara
  Participants
    Hispanic or Latino | 13 | 3 | 2 | 0 | 0 | 2 | 0 | 20
    Not Hispanic or Latino | 91 | 62 | 69 | 6 | 7 | 28 | 17 | 280
    Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 13 | 5 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants for Nivo mono, Nivo + Ipi , Nivo + Liri and all randomized participants for Nivo Dara
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Black or African American | 11 | 5 | 7 | 0 | 0 | 1 | 2 | 26
    White | 89 | 58 | 63 | 5 | 7 | 38 | 19 | 279
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 2 | 1 | 2 | 1 | 0 | 4 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Drug Related Grade 3-4 AEs
Description: Number and percent of participants that experienced drug related Grade 3-4 AEs occurring up to 100 days after the last dose of study drug.
Time Frame: Nivo Mono: approximately up to 6 years and 9 months Nivo Ipi: approximately up to 5 months Nivo Liri: approximately up to 4 years 1 month
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 105 | 65 | 72
Participants | 19 | 18 | 0

2. Primary Outcome: Number of Participants That Experienced Drug Related Grade 3-4 SAEs
Description: Number and percent of participants that experienced drug related Grade 3-4 SAEs occurring up to 100 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 105 | 65 | 72
Participants | 28 | 8 | 3

3. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities by Worst Toxicity Grade - Liver
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 105 | 65 | 72
Participants
  ALT OR AST > 3XULN: number analyzed (Participants) | 105 | 59 | 72
  ALT OR AST > 3XULN | 3 | 1 | 4
  ALT OR AST > 5XULN: number analyzed (Participants) | 105 | 59 | 72
  ALT OR AST > 5XULN | 1 | 0 | 2
  ALT OR AST > 10XULN: number analyzed (Participants) | 105 | 59 | 72
  ALT OR AST > 10XULN | 1 | 0 | 1
  ALT OR AST > 20XULN: number analyzed (Participants) | 105 | 59 | 72
  ALT OR AST > 20XULN | 1 | 0 | 0
  TOTAL BILIRUBIN > 2XULN: number analyzed (Participants) | 105 | 59 | 72
  TOTAL BILIRUBIN > 2XULN | 1 | 1 | 2
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN ONE DAY: number analyzed (Participants) | 105 | 59 | 72
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN ONE DAY | 1 | 0 | 1
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN 30 DAYS: number analyzed (Participants) | 105 | 59 | 72
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN 30 DAYS | 1 | 0 | 1

4. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities by Worst Toxicity Grade - Thyroid
Time Frame: as for outcome 1
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 83 | 47 | 72
Participants
  TSH > ULN | 14 | 19 | 15
  TSH > ULN WITH TSH <= ULN AT BASELINE | 11 | 13 | 9
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN | 0 | 7 | 1
  TSH > ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 1 | 1 | 1
  TSH > ULN WITH FT3/FT4 TEST MISSING | 13 | 11 | 13
  TSH < LLN | 8 | 6 | 6
  TSH < LLN WITH TSH >= LLN AT BASELINE | 5 | 6 | 4
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 0 | 1 | 1
  TSH < LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0 | 0 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 8 | 5 | 5

5. Primary Outcome: Number of Participants That Experienced Drug-related Grade 3-4 AEs in the Nivolumab + Daratumumab Cohort
Time Frame: approximately up to 4 years
Population: All treated participants in the nivo dara cohort
Measure: Count of Participants; unit: Participants
Groups:
- Nivolumab + Daratumumab_Cohort A1: ND Regimen
  Each cycle is 28 days
  Nivolumab:
  Cycle 1: 240 mg iv Day 15 Cycle 2-6: 240 mg iv Days 1, 15 Cycle 7 & beyond: 480 mg iv Day 1
  Daratumumab:
  Cycle 1-2: 16 mg/kg iv Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg iv Days 1, 15 Cycle 7 & beyond: 16 mg/kg iv Day 1
  Pomalidomide:
  4 mg po daily (Days 1-21) of each 28-day cycle
  Dexamethasone:
  Weeks without daratumumab dosing 40 mg po per day (Days 1, 8, 15, 22) of each 28-day cycle for subjects 75 years old 20 mg po per day (Days 1, 8, 15, 22) of each 28-day cycle for subjects > 75 years old
- Nivolumab + Daratumumab_Cohort A2: ND-Pd Regimen
  Each cycle is 28 days
  Nivolumab:
  Cycle 1: 240 mg iv Day 15 Cycle 2-6: 240 mg iv Days 1, 15 Cycle 7 & beyond: 480 mg iv Day 1
  Daratumumab:
  Cycle 1-2: 16 mg/kg iv Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg iv Days 1, 15 Cycle 7 & beyond: 16 mg/kg iv Day 1
- Nivolumab + Daratumumab_Cohort B1: ND Regimen
  Each cycle is 28 days
  Nivolumab:
  Cycle 1: 240 mg iv Day 15 Cycle 2 & beyond: 480 mg iv Day 1
  Daratumumab:
  Cycle 1*-2: 16 mg/kg iv Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg iv Days 1, 15 Cycle 7 & beyond: 16 mg/kg iv Day 1
- Nivolumab + Daratumumab_Cohort B2: D Monotherapy Regimen
  Each cycle is 28 days
  Daratumumab:
  Cycle 1*-2: 16 mg/kg iv Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg iv Days 1, 15 Cycle 7 & beyond: 16 mg/kg iv Day 1
Arm/Group | Nivolumab + Daratumumab_Cohort A1 | Nivolumab + Daratumumab_Cohort A2 | Nivolumab + Daratumumab_Cohort B1 | Nivolumab + Daratumumab_Cohort B2
Number analyzed (Participants) | 6 | 5 | 41 | 22
Participants | 2 | 5 | 13 | 2

6. Primary Outcome: Number of Participants That Experienced Drug-related Grade 3-4 SAEs in the Nivolumab + Daratumumab Cohort
Time Frame: approximately up to 4 years
Population: All treated participants in the nivo dara cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab_Cohort A1 | Nivolumab + Daratumumab_Cohort A2 | Nivolumab + Daratumumab_Cohort B1 | Nivolumab + Daratumumab_Cohort B2
Number analyzed (Participants) | 6 | 5 | 41 | 22
Participants | 2 | 4 | 10 | 6

7. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities by Worst Toxicity Grade in the Nivolumab + Daratumumab Cohort - Hematology
Time Frame: approximately up to 4 years
Population: All treated participants in the nivo dara cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab_Cohort A1 | Nivolumab + Daratumumab_Cohort A2 | Nivolumab + Daratumumab_Cohort B1 | Nivolumab + Daratumumab_Cohort B2
Number analyzed (Participants) | 6 | 5 | 41 | 22
Participants
  Hemoglobin: number analyzed (Participants) | 6 | 5 | 41 | 21
  Hemoglobin: Grade 0 | 0 | 0 | 3 | 1
  Hemoglobin: Grade 1 | 2 | 2 | 13 | 13
  Hemoglobin: Grade 2 | 2 | 2 | 20 | 5
  Hemoglobin: Grade 3 | 2 | 1 | 5 | 2
  Hemoglobin: Grade 4 | 0 | 0 | 0 | 0
  Platelet count: number analyzed (Participants) | 6 | 5 | 41 | 21
  Platelet count: Grade 0 | 3 | 1 | 19 | 8
  Platelet count: Grade 1 | 2 | 3 | 11 | 9
  Platelet count: Grade 2 | 0 | 1 | 3 | 3
  Platelet count: Grade 3 | 0 | 0 | 3 | 0
  Platelet count: Grade 4 | 1 | 0 | 5 | 1
  Leukocytes: number analyzed (Participants) | 6 | 5 | 41 | 21
  Leukocytes: Grade 0 | 2 | 0 | 10 | 5
  Leukocytes: Grade 1 | 1 | 0 | 6 | 9
  Leukocytes: Grade 2 | 2 | 2 | 15 | 5
  Leukocytes: Grade 3 | 0 | 2 | 9 | 2
  Leukocytes: Grade 4 | 1 | 1 | 1 | 0
  Lymphocytes (Absolute): number analyzed (Participants) | 6 | 5 | 41 | 21
  Lymphocytes (Absolute): Grade 0 | 3 | 0 | 6 | 3
  Lymphocytes (Absolute): Grade 1 | 0 | 0 | 9 | 5
  Lymphocytes (Absolute): Grade 2 | 0 | 0 | 9 | 7
  Lymphocytes (Absolute): Grade 3 | 2 | 3 | 15 | 5
  Lymphocytes (Absolute): Grade 4 | 1 | 2 | 2 | 1
  Absolute Neutrophil Count: Grade 0 | 3 | 0 | 14 | 10
  Absolute Neutrophil Count: Grade 1 | 2 | 0 | 8 | 6
  Absolute Neutrophil Count: Grade 2 | 0 | 0 | 6 | 6
  Absolute Neutrophil Count: Grade 3 | 1 | 3 | 9 | 0
  Absolute Neutrophil Count: Grade 4 | 0 | 2 | 4 | 0

8. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities by Worst Toxicity Grade in the Nivolumab + Daratumumab Cohort - Liver
Time Frame: approximately up to 4 years
Population: All treated participants in the nivo dara cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab_Cohort A1 | Nivolumab + Daratumumab_Cohort A2 | Nivolumab + Daratumumab_Cohort B1 | Nivolumab + Daratumumab_Cohort B2
Number analyzed (Participants) | 6 | 5 | 41 | 22
Participants
  ALT or AST >3xULN | 0 | 0 | 0 | 0
  ALT or AST >5xULN | 1 | 3 | 9 | 0
  ALT or AST >10xULN | 1 | 3 | 9 | 0
  ALT or AST >20xULN | 1 | 3 | 9 | 0
  Total Bilirubin > 2xULN | 1 | 3 | 9 | 0
  ALT or AST >3xULN with total Bilirubin > 2xULN within 1 day | 1 | 3 | 9 | 0
  ALT or AST >3xULN with total Bilirubin >2xULN within 30 days | 1 | 3 | 9 | 0

9. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities by Worst Toxicity Grade in the Nivolumab + Daratumumab Cohort - Thyroid
Time Frame: approximately up to 4 years
Population: All treated participants in the nivo dara cohort with at Least One On-Treatment TSH Measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab_Cohort A1 | Nivolumab + Daratumumab_Cohort A2 | Nivolumab + Daratumumab_Cohort B1 | Nivolumab + Daratumumab_Cohort B2
Number analyzed (Participants) | 6 | 5 | 38 | 19
Participants
  TSH>ULN | 3 | 1 | 8 | 3
  TSH > ULN WITH TSH <= ULN AT BASELINE | 1 | 1 | 7 | 2
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN (A) | 1 | 0 | 1 | 0
  TSH > ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 0 | 0 | 5 | 2
  WITH FT3/FT4 TEST MISSING | 2 | 1 | 2 | 1
  TSH < LLN | 0 | 2 | 2 | 2
  TSH < LLN WITH TSH >= LLN AT BASELINE | 0 | 2 | 2 | 1
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 0 | 0 | 0 | 0
  TSH < LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0 | 0 | 1 | 2
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 2 | 1 | 0

10. Secondary Outcome: Best Overall Response
Description: the best response designation over the study as a whole, recorded between the date of first dose and the last efficacy assessment prior to subsequent therapy.
  Measured in Complete Response and Partial Response
Time Frame: as for outcome 1
Population: All treated participants with available measurements (excluding Multiple Myeloma (MM) Group)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 77 | 58 | 62
Percentage of participants
  Complete Response | 10.4 [4.6 to 19.4] | 13.8 [6.1 to 25.4] | 9.7 [3.6 to 19.9]
  Partial Response | 33.8 [23.4 to 45.4] | 34.5 [22.5 to 48.1] | 29.0 [18.2 to 41.9]

11. Secondary Outcome: Best Overall Response - Multiple Myeloma Group
Description: the best response designation over the study as a whole, recorded between the date of first dose and the last efficacy assessment prior to subsequent therapy.
Time Frame: as for outcome 1
Population: All Treated participants with available measurements in the Multiple Myeloma (MM) Group
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 27 | 7 | 10
Percentage
  Complete Remission | 3.7 [0.1 to 19.0] | 0 [0.0 to 41.0] | 0 [0.0 to 30.8]
  Partial Remission | 0 [0.0 to 12.8] | 0 [0.0 to 41.0] | 0 [0.0 to 30.8]
  Very Good Partial Response: number analyzed (Participants) | 27 | 7 | 0
  Very Good Partial Response | 0 [0.0 to 12.8] | 0 [0.0 to 41.0] |
  Stringent Compete Response: number analyzed (Participants) | 27 | 7 | 0
  Stringent Compete Response | 0 [0.0 to 12.8] | 0 [0 to 41.0] |

12. Secondary Outcome: Duration of Response
Description: the best response designation over the study as a whole, recorded between the date of first dose and the last efficacy assessment prior to subsequent therapy.
  Measured in Complete Remission and Partial Remission
Time Frame: Nivo Mono: approximately up to 6 years and 9 months Nivo Ipi: approximately up to approximately 37 months Nivo Liri: approximately up to 4 years 1 month
Population: All Responding participants (Complete Response and Partial Response) with available measurements (excluding Multiple Myeloma (MM) Group)
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 34 | 28 | 24
Months | 22.83 [0.0 to 48.6] | 24.84 [0.0 to 36.5] | 19.38 [0.0 to 45.5]

13. Secondary Outcome: Duration of Response - Multiple Myeloma Group
Description: as for outcome 10
Time Frame: as for outcome 1
Population: All Responding participants (Complete Response and Partial Response) in the Multiple Myeloma (MM) Group
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 1 | 0 | 0
Months | NA [NA to NA] — Median value and Full Range could not be determined because of a single participant analyzed |  |

14. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) is defined as the time between date of randomization and date of progression or death, whichever occurs first. Participants who died without a reported prior progression were considered to have progressed on the date of their death. Subjects who did not progress or die were censored on the date of their last efficacy assessment.
Time Frame: From date of randomization to date of progression or death, whichever occurs first (up to approximately 24 months)
Population: All Treated Participants with available measurements
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 104 | 65 | 72
Months | 6.24 [3.48 to 9.79] | 6.93 [2.79 to 19.15] | 3.02 [1.84 to 5.52]

15. Secondary Outcome: Progression Free Survival Rate
Description: The percentage of participants remaining progression free at the specified timepoints (up to 48 Months)
Time Frame: From randomization to the specified timepoints (up to 48 months)
Population: All Treated Participants with available measurements
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 104 | 65 | 72
Percentage of Participants
  2 Months: number analyzed (Participants) | 0 | 0 | 72
  2 Months |  |  | 58.0 [45.3 to 68.8]
  4 Months: number analyzed (Participants) | 0 | 0 | 72
  4 Months |  |  | 42.4 [30.4 to 54.0]
  6 Months | 50.5 [39.8 to 60.3] | 51.5 [38.1 to 63.4] | 34.3 [23.0 to 45.8]
  9 Months: number analyzed (Participants) | 0 | 0 | 72
  9 Months |  |  | 32.5 [21.4 to 44.0]
  12 Months: number analyzed (Participants) | 104 | 65 | 0
  12 Months | 34.8 [24.2 to 45.5] | 45.3 [32.0 to 57.7] |
  18 Months: number analyzed (Participants) | 104 | 65 | 0
  18 Months | 31.0 [20.7 to 42.0] | 40.1 [26.8 to 53.1] |
  24 Months: number analyzed (Participants) | 104 | 65 | 0
  24 Months | 20.3 [11.1 to 31.5] | 30.9 [18.0 to 44.9] |
  36 Months: number analyzed (Participants) | 104 | 0 | 0
  36 Months | 15.8 [7.6 to 26.8] |  |
  48 Months: number analyzed (Participants) | 104 | 0 | 0
  48 Months | 13.2 [5.6 to 24.1] |  |

16. Secondary Outcome: Overall Survival
Description: The percentage of participants remaining alive. Median values are computed using Kaplan-Meier method
Time Frame: Nivo Mono: approximately up to 6 years and 9 months Nivo Ipi: approximately up to3 years Nivo Liri: approximately up to 4 years 1 month
Population: All Treated Participants with available measurements
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 104 | 65 | 72
Months | 52.57 [29.0 to NA] — Upper limit number not reached | 30.39 [13.24 to NA] — upper limit number not reached | 14.95 [9.36 to 34.23]

17. Secondary Outcome: Number of Participants With PD-L1 Expression
Description: Number of Participants with PD-L1 expression in the following categories
  * baseline PD-L1 expression ≥ 1%
  * baseline PD-L1 expression < 1%
  * without PD-L1 quantifiable at baseline
Time Frame: At baseline (prior to start of study treatment)
Population: All Treated Participants
Measure: Number; unit: Number of Participants
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 105 | 65 | 72
Number of Participants
  Baseline PD-L1 expression ≥ 1% | 25 | 26 | 16
  Baseline PD-L1 expression < 1% | 16 | 14 | 20
  PD-L1 not quantifiable at baseline | 64 | 25 | 36

18. Secondary Outcome: Percentage Change From Baseline in the Modified Severity Weighted Assessment Tool (mSWAT) Score
Description: mSWAT is a scoring technique involving the direct assessment of the percentage of body-surface-area (BSA) affected by skin lesions.
  There are 12 body regions (each one assigned a different percentage of BSA). For each body region, the assigned BSA percentage is multiplied by a factor weighing the type and severity of lesion observed (patch= x1, plaque = x2, tumor= x4).
  The sum of the individual body region sub-scores is then summed to generate the final mSWAT score, which ranges from 0 (best outcome) to 400 (worst outcome).
Time Frame: From baseline (last measurement before start of study treatment) to last available measurement after start of study treatment (88 weeks for Nivo mono, 93 weeks for nivo+ipi, 25 weeks for nivo+liri)
Population: All Treated Participants with cutaneous T Cell lymphoma and available measurements
Measure: Mean (Standard Deviation); unit: Percent of change from baseline
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab
Number analyzed (Participants) | 1 | 1 | 1
Percent of change from baseline | 8.70 (NA) — Only 1 participant with available measurements at baseline and 88 weeks | 63.03 (NA) — Only 1 participant with available measurements at baseline and 93 weeks | -39.49 (NA) — Only 1 participant with available measurements at baseline and 25 weeks

19. Secondary Outcome: Time to MRD Negativity Status in the Nivolumab + Daratumumab Cohort
Description: Time to MRD Negativity status in specific NGS and NGF sensitivity levels
Time Frame: approximately up to 4 years
Population: All Randomized MRD Evaluable Subjects Achieving MRD Negativity
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Cohort A-1: ND Regimen
  Each cycle is 28 days
  Nivolumab:
  Cycle 1: 240 mg iv Day 15 Cycle 2-6: 240 mg iv Days 1, 15 Cycle 7 & beyond: 480 mg iv Day 1
  Daratumumab:
  Cycle 1-2: 16 mg/kg iv Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg iv Days 1, 15 Cycle 7 & beyond: 16 mg/kg iv Day 1
  Pomalidomide:
  4 mg po daily (Days 1-21) of each 28-day cycle
  Dexamethasone:
  Weeks without daratumumab dosing 40 mg po per day (Days 1, 8, 15, 22) of each 28-day cycle for subjects 75 years old 20 mg po per day (Days 1, 8, 15, 22) of each 28-day cycle for subjects > 75 years old
- Cohort A-2: ND-Pd Regimen
  Each cycle is 28 days
  Nivolumab:
  Cycle 1: 240 mg iv Day 15 Cycle 2-6: 240 mg iv Days 1, 15 Cycle 7 & beyond: 480 mg iv Day 1
  Daratumumab:
  Cycle 1-2: 16 mg/kg iv Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg iv Days 1, 15 Cycle 7 & beyond: 16 mg/kg iv Day 1
- Cohort B-1: ND Regimen
  Each cycle is 28 days
  Nivolumab:
  Cycle 1: 240 mg iv Day 15 Cycle 2 & beyond: 480 mg iv Day 1
  Daratumumab:
  Cycle 1*-2: 16 mg/kg iv Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg iv Days 1, 15 Cycle 7 & beyond: 16 mg/kg iv Day 1
- Cohort B-2: D Monotherapy Regimen
  Each cycle is 28 days
  Daratumumab:
  Cycle 1*-2: 16 mg/kg iv Days 1, 8, 15, 22 Cycle 3-6: 16 mg/kg iv Days 1, 15 Cycle 7 & beyond: 16 mg/kg iv Day 1
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 1 | 0 | 6 | 4
Months
  NGS sensitivity level=10e-4: number analyzed (Participants) | 1 | 0 | 6 | 1
  NGS sensitivity level=10e-4 | 3.02 (NA) — SD not calculable with 1 participant |  | 3.60 (2.409) | 2.83 (NA) — SD not calculable with 1 participant
  NGS sensitivity level=10e-5: number analyzed (Participants) | 1 | 0 | 6 | 0
  NGS sensitivity level=10e-5 | 3.02 (NA) — SD not calculable with 1 participant |  | 5.45 (4.788) |
  NGS sensitivity level=10e-6: number analyzed (Participants) | 1 | 0 | 0 | 0
  NGS sensitivity level=10e-6 | 30.85 (NA) — SD not calculable with 1 participant |  |  |
  NGF sensitivity level=10e-4: number analyzed (Participants) | 0 | 0 | 4 | 4
  NGF sensitivity level=10e-4 |  |  | 2.94 (0.230) | 4.20 (2.766)
  NGF sensitivity level=10e-5: number analyzed (Participants) | 0 | 0 | 3 | 0
  NGF sensitivity level=10e-5 |  |  | 6.97 (6.776) |
  NGF sensitivity level=10e-6: number analyzed (Participants) | 0 | 0 | 2 | 0
  NGF sensitivity level=10e-6 |  |  | 12.30 (3.508) |

20. Secondary Outcome: Objective Response Rate in the Nivolumab + Daratumumab Cohort
Time Frame: approximately up to 4 years
Population: All randomized participants in the nivo dara cohort
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 6 | 7 | 43 | 22
Percentage | 66.7 [22.3 to 95.7] | 71.4 [29.0 to 93.3] | 51.2 [35.5 to 66.7] | 36.4 [17.2 to 59.3]

21. Secondary Outcome: Duration of Response in the Nivolumab + Daratumumab Cohort
Time Frame: approximately up to 4 years
Population: All randomized participants in the nivo dara cohort
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 6 | 7 | 43 | 22
Months | NA [6.47 to NA] — inusufficient number of participants with a response to calculable by KM methodology | NA [9.30 to NA] — inusufficient number of participants with a response to calculable by KM methodology | 6.70 [3.71 to 14.29] | 12.98 [2.20 to NA] — inusufficient number of participants with a response to calculable by KM methodology

22. Secondary Outcome: Progression Free Survival in the Nivolumab + Daratumumab Cohort
Time Frame: approximately up to 4 years
Population: All randomized participants in the nivo dara cohort
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 6 | 7 | 43 | 22
Months | 7.56 [3.19 to NA] — Insufficient number of events to calculate via KM methodology | 16.95 [NA to NA] — Insufficient number of events to calculate via KM methodology | 7.49 [4.67 to 9.46] | 7.01 [2.96 to 12.94]

23. Secondary Outcome: Cmax in the Nivolumab + Daratumumab Cohort
Description: Maximum observed serum concentration
Time Frame: approximately up to 4 years
Population: All treated participants - Please note that blood sampling collection for PK endpoints was limited to end-of-infusion samples and pre-dose samples only. Because there was no blood sampling throughout a dosing interval, values for this PK endpoint can't be determined as we do not have the raw nivolumab concentration-time data necessary to do so. Hence, number of participants analyzed is set at 0
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Tmax in the Nivolumab + Daratumumab Cohort
Description: Time of maximum observed serum concentration
Time Frame: approximately up to 4 years
Population: as for outcome 23
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Secondary Outcome: Cmin in the Nivolumab + Daratumumab Cohort
Description: Serum concentration achieved at the end of dosing interval (trough concentration)
Time Frame: approximately up to 4 years
Population: as for outcome 23
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: AUC (0-T) in the Nivolumab + Daratumumab Cohort
Description: Area under the plasma concentration-time curve from time zero to the last time of the last quantifiable concentration
Time Frame: approximately up to 4 years
Population: as for outcome 23
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

27. Secondary Outcome: AUC (TAU) in the Nivolumab + Daratumumab Cohort
Description: Area under the concentration-time curve in one dosing interval
Time Frame: approximately up to 4 years
Population: as for outcome 23
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

28. Secondary Outcome: End of Infusion Nivolumab Concentration Levels in the Nivolumab + Daratumumab Cohort
Description: Serum concentration achieved at the end of study drug infusion
Time Frame: Measurements collected at cycles 1, 2, 3, 5, 7, and 11; each cycle is 28 days
Population: All treated participants in the nivo dara cohort - pharmacokinetic subset
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort A-1 | Cohort A-2 | Cohort B-1 | Cohort B-2
Number analyzed (Participants) | 6 | 5 | 41 | 0
ug/mL
  Cycle 1: number analyzed (Participants) | 5 | 0 | 32 | 0
  Cycle 1 | 57.28 (6.78) |  | 69.59 (18.79) |
  Cycle 2: number analyzed (Participants) | 0 | 0 | 21 | 0
  Cycle 2 |  |  | 175.73 (88.94) |
  Cycle 3: number analyzed (Participants) | 5 | 0 | 6 | 0
  Cycle 3 | 105.14 (31.41) |  | 193.38 (69.74) |
  Cycle 5: number analyzed (Participants) | 0 | 0 | 21 | 0
  Cycle 5 |  |  | 208.14 (58.38) |
  Cycle 7: number analyzed (Participants) | 4 | 1 | 3 | 0
  Cycle 7 | 227.75 (26.79) | 206.00 (NA) — Not calculable with only 1 participant | 193.00 (70.06) |
  Cycle 11: number analyzed (Participants) | 0 | 1 | 3 | 0
  Cycle 11 |  | 206.00 (NA) — Not calculable with only 1 participant | 212.00 (38.20) |

ADVERSE EVENTS:
Time Frame: Nivo Mono: approximately up to 6 years and 9 months Nivo Ipi: approximately up to 5 months Nivo Liri: approximately up to 4 years 1 month Nivo Dara: approximately 4 years
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Nivolumab + Daratumumab Cohort A1: ND regimen: Nivolumab (240 mg up to cycle 6, then 480 mg) + Daratumumab (16 mg/Kg)
Arm/Group | Nivolumab Monotherapy (Expansion) | Nivolumab + Ipilimumab | Nivolumab + Lirilumab | Nivolumab + Daratumumab Cohort A1 | Nivolumab + Daratumumab_Cohort A2 | Nivolumab + Daratumumab_Cohort B1 | Nivolumab + Daratumumab_Cohort B2
All-Cause Mortality (participants affected / at risk) | 53/105 | 33/65 | 42/72 | 1/6 | 3/7 | 24/42 | 13/23
Serious Adverse Events (participants affected / at risk) | 50/105 | 39/65 | 34/72 | 3/6 | 5/5 | 15/41 | 9/22
Other Adverse Events (participants affected / at risk) | 102/105 | 62/65 | 69/72 | 6/6 | 5/5 | 35/41 | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Monotherapy (Expansion) (N=105) | Nivolumab + Ipilimumab (N=65) | Nivolumab + Lirilumab (N=72) | Nivolumab + Daratumumab Cohort A1 (N=6) | Nivolumab + Daratumumab_Cohort A2 (N=5) | Nivolumab + Daratumumab_Cohort B1 (N=41) | Nivolumab + Daratumumab_Cohort B2 (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 6 | 7 | 1 | 0 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 3 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 5 | 2 | 2 | 2 | 1 | 3
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 13 | 14 | 1 | 0 | 3 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 4 | 0 | 0 | 0 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fistula of small intestine (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 4 | 2 | 2 | 0 | 0 | 0 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 3 | 3 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome with single lineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Stent malfunction (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 3 | 3 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Monotherapy (Expansion) (N=105) | Nivolumab + Ipilimumab (N=65) | Nivolumab + Lirilumab (N=72) | Nivolumab + Daratumumab Cohort A1 (N=6) | Nivolumab + Daratumumab_Cohort A2 (N=5) | Nivolumab + Daratumumab_Cohort B1 (N=41) | Nivolumab + Daratumumab_Cohort B2 (N=22)
Anaemia (Blood and lymphatic system disorders) | 23 | 12 | 18 | 3 | 4 | 10 | 4
Neutropenia (Blood and lymphatic system disorders) | 12 | 6 | 7 | 1 | 4 | 9 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 7 | 5 | 1 | 1 | 5 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 7 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 6 | 10 | 1 | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 4 | 4 | 0 | 2 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 10 | 5 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 12 | 10 | 15 | 0 | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 28 | 20 | 21 | 1 | 4 | 6 | 4
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 2 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 24 | 17 | 15 | 1 | 2 | 4 | 2
Vomiting (Gastrointestinal disorders) | 13 | 9 | 8 | 1 | 2 | 2 | 0
Asthenia (General disorders) | 3 | 3 | 3 | 0 | 1 | 4 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 10 | 10 | 6 | 0 | 1 | 0 | 2
Fatigue (General disorders) | 46 | 30 | 30 | 2 | 2 | 8 | 3
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 4 | 0 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 3 | 4 | 4 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 11 | 8 | 7 | 1 | 2 | 1 | 1
Pain (General disorders) | 5 | 4 | 3 | 0 | 0 | 3 | 0
Peripheral swelling (General disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 27 | 25 | 8 | 1 | 1 | 4 | 3
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 5 | 1
Bronchitis haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 4 | 1 | 0 | 3 | 3 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 6 | 4 | 1 | 1 | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 17 | 10 | 13 | 2 | 4 | 9 | 3
Urinary tract infection (Infections and infestations) | 7 | 4 | 3 | 0 | 0 | 2 | 2
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0 | 1 | 3 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 10 | 13 | 2 | 2 | 10 | 4
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 5 | 4 | 0 | 2 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 7 | 6 | 1 | 0 | 3 | 0
Blood bilirubin increased (Investigations) | 2 | 4 | 3 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 10 | 3 | 4 | 1 | 0 | 2 | 3
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Lipase increased (Investigations) | 9 | 8 | 3 | 1 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 6 | 0 | 3 | 2 | 0
Platelet count decreased (Investigations) | 0 | 2 | 7 | 0 | 2 | 0 | 1
White blood cell count decreased (Investigations) | 4 | 4 | 8 | 0 | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 17 | 12 | 14 | 0 | 1 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 6 | 2 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 9 | 4 | 4 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 11 | 8 | 1 | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4 | 3 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 12 | 3 | 2 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 14 | 7 | 5 | 1 | 0 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 3 | 1 | 0 | 1 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0 | 4 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 5 | 7 | 0 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 5 | 5 | 0 | 1 | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 10 | 11 | 3 | 3 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 11 | 14 | 0 | 1 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 1 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 3 | 0 | 2 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 3 | 1 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5 | 1 | 2 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3 | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 5 | 6 | 1 | 1 | 3 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 2 | 2 | 0 | 2 | 3 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 16 | 7 | 5 | 0 | 3 | 3 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3 | 1 | 1 | 1 | 3 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 7 | 10 | 5 | 1 | 0 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 3 | 1 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 22 | 11 | 3 | 2 | 4 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 7 | 2 | 3 | 5 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 4 | 2 | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 2 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 3 | 2 | 1 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 2 | 2 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 11 | 9 | 1 | 4 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 22 | 12 | 8 | 0 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 8 | 5 | 0 | 0 | 3 | 1
Flushing (Vascular disorders) | 3 | 0 | 0 | 0 | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 5 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 6 | 1 | 1 | 0 | 0 | 3 | 1
Hypotension (Vascular disorders) | 8 | 1 | 3 | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 13 | 1 | 4 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 9 | 2 | 1 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 2 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 4 | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 11 | 9 | 8 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 13 | 8 | 5 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 6 | 9 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 6 | 9 | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 6 | 4 | 2 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 4 | 7 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 | 6 | 2 | 0 | 0 | 0 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 4 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 9 | 2 | 1 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 6 | 2 | 5 | 0 | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 2 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 1 | 4 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 4 | 4 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT01592370/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT01592370/SAP_001.pdf